CLINICAL TRIAL: NCT05864859
Title: Investigation of the Effect of Birth Experience With a Wearable Simulated Motherhood Model on Empathic Tendency and Privacy Protection Level: A Randomized Controlled Study
Brief Title: Empathic Tendency and Privacy Protection Level
Acronym: SCIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KaratayUNIH3
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-05

CONDITIONS: Simulation; Empathy
Keywords: Simulation; Empathy; Privacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal birth group (Experimental): It consisted of preliminary information (10 minutes), practice (10 minutes) and analysis (20 minutes) sessions with groups of 2 people (1 midwife, 1 pregnant) accompanied by a scenario where there was no complication during labor.
  Interventions: Other: Simulation
- Breech birth group (Experimental): It consisted of preliminary information (10 minutes), practice (10 minutes) and analysis (20 minutes) sessions with groups of 2 people (1 midwife, 1 pregnant) accompanied by a scenario that experienced complications during labor.
  Interventions: Other: Simulation
- Control group (No Intervention): She continued her education in accordance with the (1+32) hour curriculum within the scope of the midwifery undergraduate program Integrated Practice I and EBE402 Integrated Practice II courses.

INTERVENTIONS:
Other: Simulation — In the simulation session, while 2 participants (1 midwife, 1 pregnant) performed the roles in accordance with the clinical scenario, the performance was recorded in the control room. A Wearable Pregnancy Simulator was worn by the student performing the pregnant role. During the simulation, the participants were able to interact with the facilitators when they had questions. The application time did not exceed 10 minutes.
  Arms: Breech birth group; Normal birth group

SUMMARY:
Proving the empathy level and privacy protection effectiveness of the low-cost, high-reality and interactive education model constitutes the original value of the project and our main motivation. The project has a unique value for a sustainable future in terms of its impact at the social level in terms of midwifery students in particular and positive birth experience and qualified midwifery care in general. It will also provide data for the comparison of innovative education methods with traditional education methods. Thus, it will help to improve, regulate or build capacity of future initiatives.

DETAILED DESCRIPTION:
Humanistic care is also conceptualized as the ability to communicate with patients, feel their emotions, meet their needs, and develop harmonious therapeutic relationships. Humanistic care is the essence and connotation of the care process. But developing a sense of humanistic care is quite difficult. Despite emphasizing humanistic care in midwifery education and making great efforts, its integration into professional practice is still not at the desired level .

Empathy refers to the tendency to recognize, help, and respond to other people's experiences and emotions. Empathy allows midwives to measure various situations, understand mothers' situation, perspective, feelings, and apply appropriate woman-centered care. It is stated that empathy can contribute to students' humanistic care skills both directly and indirectly through emotional intelligence.

Birth is one of the most private areas where privacy should be protected, and practices done during childbirth cause embarrassment in women, decrease the level of satisfaction and lead to a negative perception of childbirth. Healthcare professionals have both ethical and legal responsibilities regarding privacy. In order to fulfill their duties towards the individuals they care for, they need to protect the privacy of the individual. In a meta-analysis study examining the ethical decision-making process in care and practices, it was found that it is a difficult process to implement the ethical decision-making process and it is affected by many personal and situational factors.

The use of standardized patient or human actors in simulation practice was initiated in 1963 by a neurologist from the University of Southern California. It is stated that the use of standardized patient or human actors adds more realism to the simulation by allowing training in both procedural and communication skills. With the hybrid simulation, which allows the birth process to be animated as in real life, the human element in birth is preserved and the reality shock they will experience in real life is prevented. It is stated that it adds more realism and interaction thanks to psychological reactions, especially during a clinical event.

It is stated that the use of simulation reflection, role playing, pedagogical theater and real-life case studies should be included in the curriculum in midwifery programs. However, it is stated that there are limited studies with midwifery students. It is stated that the use of standardized patients is beneficial not only for learners, but also for standardized patients themselves. Therefore, it is suggested that more research is needed to examine the mutual benefits of using standardized patients in simulation practice. In this context, proving the empathy level and privacy protection effectiveness of the low-cost, high-reality and interactive education model in line with the literature proposal constitutes the original value of the project and our main motivation. The project has a unique value for a sustainable future in terms of its impact at the social level in terms of midwifery students in particular and positive birth experience and qualified midwifery care in general. It will also provide data for the comparison of innovative education methods with traditional education methods. Thus, it will help to improve, regulate or build capacity of future initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Being a final year midwifery student,
* Not being married
* To be nulliparous
* Volunteering to participate in research

Exclusion Criteria:

* Having the ability to read, listen, write, speak and understand Turkish,
* Repeating the course,
* Unwilling to withdraw from research

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Privacy | 1 years
  Privacy Protection Scale in Obstetrics and Gynecology: The scale has 2 sections: awareness level and application frequency, 2 sub-dimensions: physical-social privacy (items 1-15) and psychological-information privacy (items 16-30) and the total It consists of 30 items. There are no items that need to be reversed in calculating the total scale score. The Cronbach Alpha reliability coefficient of the scale is 0.95 for the level of awareness section, 0.96 for the frequency of application section, 0.90 and 0.92 for the physical-social privacy sub-dimension, and 0.93 and 0.94 for the psychological-information privacy sub-dimension. was found as. The increase in the scores individuals receive from the scale indicates that their privacy awareness levels are high and their frequency of privacy-oriented practices is high.A minimum score of 30 and a maximum score of 150 is obtained from the scale.
Empathy | 1 years
  Empathic Tendency Scale (EES): Empathic Tendency A validity and reliability study of the scale was conducted and the reliability coefficient was found to be 0.82. This is what was done In the study, the Cronbach alpha coefficient was determined as 0.75. Individuals express their agreement with the opinion in the relevant article by marking one of the numbers from 1 to 5 next to each item. The marked numbers constitute the scores for that item. The highest total score that can be obtained is 100 and the lowest score is 20. A high total score means that the empathic tendency is high. Some expressions in the empathic tendency scale are written negatively and reversed to prevent people from saying "yes". To avoid the tendency to say yes, the statements in the 3rd, 6th, 7th, 8th, 11th, 12th, 13th, 15th rows are written backwards. The scoring for these items is; It was determined as completely inappropriate (5 points) and completely appropriate (1 point).

CONTACTS AND LOCATIONS:
Overall Officials: Hediye KARAKOÇ, Study Chair — KTO Karatay University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakoc H, Ozkan H. The effect of wearable simulated birth model on students' empathy and privacy protection levels: a randomised controlled trial. BMC Med Educ. 2026 Feb 5. doi: 10.1186/s12909-025-08441-8. Online ahead of print. PMID 41639700